CLINICAL TRIAL: NCT07089732
Title: Evaluation of the Effects of GLP-1 Formula Liquid Drink on Gut Microbiota Modulation and Blood Glucose Regulation in Prediabetic Populations
Brief Title: Effects of a GLP-1 Formula Drink on Gut Microbiota and Glycemic Control in Prediabetic Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS2-24199
Record Dates: First submitted 2025-07-25; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Prediabetes
MeSH Terms: conditions — Obesity; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLP-1 formula liquid drink (Experimental): GLP-1 formula liquid drink, 50 g/glass jar
  Interventions: Dietary Supplement: GLP-1 formula liquid drink
- placebo (Placebo Comparator): The placebo contained the same base ingredients as the GLP-1 FORMULA but without the active GLP-1 FORMULA component.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GLP-1 formula liquid drink — One glass jar (50 g) of the GLP-1 formula liquid drink was administered once daily, 30 minutes prior to the first meal of the day.
  Arms: GLP-1 formula liquid drink
Dietary Supplement: Placebo — One glass jar (50 g) of the placebo liquid drink was administered once daily, 30 minutes prior to the first meal of the day.
  Arms: placebo

SUMMARY:
A clinical human dietary intervention trial was conducted to investigate the effects of GLP-1 FORMUL liquid supplementation in individuals with prediabetes or obesity, with a focus on improvements in glycemic and lipid parameters, body composition, and gut microbiota profiles.

DETAILED DESCRIPTION:
This 12-week randomized, placebo-controlled clinical trial aims to evaluate the nutritional and metabolic effects of GLP-1 FORMULA liquid supplementation. A total of 100 adult participants will be recruited and randomly assigned to one of two groups: (1) placebo group (n = 50), and (2) GLP-1 FORMULA group (n = 50). Participants will consume one bottle (50 g) of either GLP-1 FORMULA or placebo 30 minutes prior to their first meal each day for 8 weeks, followed by a 4-week post-intervention observation period.

Throughout the study, participants will undergo nutritional assessments including body composition analysis, waist-to-hip ratio measurements, appetite rating scales, gastrointestinal symptom questionnaires, and the Patient Health Questionnaire. Additionally, oral glucose tolerance tests (OGTT), standard blood biochemistry analyses, and fecal sample collection will be conducted at designated time points to evaluate glycemic control, metabolic markers, and gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years.
* Clinically diagnosed with prediabetes (fasting plasma glucose: 100-125 mg/dL or HbA1c: 5.7-6.4%) or with a body mass index (BMI) of 25-34.9 kg/m², male or female.
* Have not participated in similar clinical studies within the past three months.
* Able to comprehend the informed consent form, including the study procedures, potential risks, and benefits, and able to provide written informed consent.

Exclusion Criteria:

* Diagnosed with autoimmune diseases or cancer.
* Diagnosed with gastrointestinal chronic diseases such as irritable bowel syndrome, inflammatory bowel disease, Crohn's disease, celiac disease, bowel control disorders, fecal incontinence, pancreatitis, peptic ulcer disease, colorectal cancer, short bowel syndrome, ulcerative colitis, lactose intolerance, or chronic diarrhea.
* History of gastrointestinal surgery.
* Planning pregnancy in the near future (including male partners), currently pregnant, or breastfeeding women.
* Known allergy or hypersensitivity to probiotics or any of the study product ingredients.
* History of major psychiatric disorders.
* History of substance abuse or alcohol dependency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in BMI at weeks 8 and 12 | Week 0, 8 and 12
  Assessment of changes in BMI at baseline, week 8, and week 12

SECONDARY OUTCOMES:
Change from baseline in blood glucose at weeks 8 and 12 | Week 0, 8 and 12
  Assessment of blood glucose changes at weeks 0, 8, and 12

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan